CLINICAL TRIAL: NCT00299624
Title: Identifying Morphological and Biological Biomarkers of the Venous Thromboembolic Risk Risk Related to Aging
Brief Title: Effect of Aging on Haemostasis Parameters
Status: Completed | Type: Observational
Sponsor: Hopital Lariboisière (Other)
Responsible Party: Pr Isabelle MAHE, Hopital Lariboisière
Other Study IDs: TAPH
Record Dates: First submitted 2006-03-06; First posted 2006-03-07 (Estimated); Last update posted 2010-09-14 (Estimated); Status verified 2010-09

CONDITIONS: Aging
Keywords: venous thromboembolism risk,; elderly,; hypercoagulability; fibrinolysis; microparticles
MeSH Terms: conditions — Thrombophilia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Aging is an independent risk factor, without any clear explanation. The primary aim of the study is to depict the effect of aging on the coagulation fibrinolysis parameters and microparticles.

DETAILED DESCRIPTION:
Patients older than 40, without any acute disease and not receiving any antiaggregant and anticoagulant therapy will be included in the study. Blood tests will be performed for coagulation, fibrinolysis and microparticles measurement.

ELIGIBILITY:
Inclusion Criteria:

* age <40 2 groups : 1 : no history of VTE 2 : history of VTE

Exclusion Criteria:

* antiaggregant or anticoagulant therapy at curative dose
* arterial or thrombotic event in the last month

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Stable patients without overt acute clinical event, not receiving antiplatelet or anticoagulant treatment
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2005-10; Primary Completion 2006-08 (Actual); Study Completion 2006-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: isabelle mahé, MD PhD, Principal Investigator — MCU-PH
Locations (2):
- France (2):
  - Hopital Lariboisiere, Paris
  - Hopital Lariboisière, Paris